CLINICAL TRIAL: NCT03941288
Title: Pharmacodynamics, Pharmacogenetics, Clinical Efficacy and Safety of Cannabidiol for Gastroparesis and Functional Dyspepsia
Brief Title: Efficacy and Safety of Cannabidiol for Gastroparesis and Functional Dyspepsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-002483; R01DK122280 (NIH)
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Gastroparesis; Dyspepsia
MeSH Terms: conditions — Gastroparesis; Dyspepsia | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pharmacodynamics and clinical effects of cannabidiol (Active Comparator): Cannabidiol will be administered orally twice daily in equally divided doses starting at 2.5mg/kg per day and increasing by 2.5 to 5.0mg/kg every other day until the target dose of 20mg/kg is reached.
  Cannabidiol and the matching placebo solution (excipients alone) will be provided in identical 100ml amber glass bottles. At the end of the treatment period, the treatment solutions will be tapered (10% volume each day) over 10 days.
  Interventions: Drug: Cannabidiol
- pharmacodynamics and clinical effects of placebo (Placebo Comparator): Placebo will be administered orally twice daily in equally divided doses starting at 2.5mg/kg per day and increasing by 2.5 to 5.0mg/kg every other day until the target dose of 20mg/kg is reached.
  Cannabidiol and the matching placebo solution (excipients alone) will be provided in identical 100ml amber glass bottles. At the end of the treatment period, the treatment solutions will be tapered (10% volume each day) over 10 days.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol and the matching placebo solution (excipients alone) will be provided in identical 100ml amber glass bottles. At the end of the treatment period, the treatment solutions will be tapered (10% volume each day) over 10 days.
  In accordance with Food and Drug Administration guidance, prior to starting treatment and at end of 1 month treatment, we shall obtain serum transaminases (alanine and aspartate) and total bilirubin levels. These tests will also be performed if patient develops clinical signs or symptoms suggestive of hepatic dysfunction (e.g., unexplained nausea, vomiting, right upper quadrant abdominal pain, fatigue, anorexia, or jaundice and/or dark urine); if such features develop the treatment will be interrupted or discontinued.
  Arms: Pharmacodynamics and clinical effects of cannabidiol
Other: placebo — Cannabidiol and the matching placebo solution (excipients alone) will be provided in identical 100ml amber glass bottles. At the end of the treatment period, the treatment solutions will be tapered (10% volume each day) over 10 days.
  In accordance with Food and Drug Administration guidance, prior to starting treatment and at end of 1 month treatment, we shall obtain serum transaminases (alanine and aspartate) and total bilirubin levels. These tests will also be performed if patient develops clinical signs or symptoms suggestive of hepatic dysfunction (e.g., unexplained nausea, vomiting, right upper quadrant abdominal pain, fatigue, anorexia, or jaundice and/or dark urine); if such features develop the treatment will be interrupted or discontinued.
  Arms: pharmacodynamics and clinical effects of placebo

SUMMARY:
Researchers are looking at the effects of a cannabidiol medication on stomach function in people with gastroparesis (a paralyzed stomach) and people with dyspepsia (an upset stomach caused by improper functioning of the stomach's muscles or nerves).

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastroparesis or functional dyspepsia (FD)
* Age 18-70 years
* Patients will be identified from among Mayo Clinic patients.
* Patients will have symptoms consistent with gastroparesis based on a national guideline for gastroparesis (symptoms plus delayed gastric emptying of solids). Patients with Rome IV criteria for postprandial distress syndrome (a subset of functional dyspepsia) will be selected based on gastric emptying of solids which is NOT delayed, in addition to standard FD criteria:

  * Symptoms fulfilled for the last 3 months with onset greater than 6 months before diagnosis:
  * One or more symptoms being bothersome: postprandial fullness, early satiation, epigastric pain or burning
  * Must include one or both of the following at least 3 days per week: bothersome postprandial fullness (i.e., severe enough to impact on usual activities) or bothersome early satiation (i.e., severe enough to prevent finishing a regular-size meal)
  * No evidence of organic, systemic, or metabolic disease to explain the symptoms on routine investigations.
  * Participants will have previously undergone test of gastric emptying of solids using the standardized Mayo Clinic scintigraphic method
* Ability to provide informed consent
* Absence of other diseases (structural or metabolic) which could interfere with interpretation of the study results
* Body mass index of 18-35 kg/m2
* Several medication classes, particularly those affecting gastrointestinal transit or motor functions, will be excluded, including GLP-1 receptor or amylin agonists in patients with diabetes mellitus. Stable doses of thyroid replacement, estrogen replacement, low-dose aspirin for cardioprotection, and birth control (but with adequate backup contraception, as drug interactions with birth control have not been conducted for secretin PAM) are

Exclusion Criteria:

* Patients with current H. pylori infection will be excluded.
* Pregnancy or lactation
* Rapid metabolizers for CYP3A4 or CYP2C19 [estimated prevalence of 17% and 18% respectively
* based on literature review will be excluded since this could impact assessment of effects of cannabidiol
* Patients with abnormal baseline liver transaminases (any value above UNL), since up to 3-fold, dose-related elevations of liver transaminases (ALT and/or AST) occur in 13% of treated patients (vs. 1% placebo);
* Hypersensitivity to cannabidiol or any of the ingredients in EPIDIOLEX
* Concomitant use of valproate, central nervous system (CNS) depressants and alcohol, other hepatotoxic drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2023-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng T, BouSaba J, Taylor A, Dilmaghani S, Busciglio I, Carlson P, Torres M, Ryks M, Burton D, Harmsen WS, Camilleri M. A Randomized, Controlled Trial of Efficacy and Safety of Cannabidiol in Idiopathic and Diabetic Gastroparesis. Clin Gastroenterol Hepatol. 2023 Dec;21(13):3405-3414.e4. doi: 10.1016/j.cgh.2023.07.008. Epub 2023 Jul 22. PMID 37482172
- [Derived] Atieh J, Maselli D, Breen-Lyles M, Torres M, Katzka D, Ryks M, Busciglio I, Burton D, Carlson P, Harmsen WS, Camilleri M. Cannabidiol for Functional Dyspepsia With Normal Gastric Emptying: A Randomized Controlled Trial. Am J Gastroenterol. 2022 Aug 1;117(8):1296-1304. doi: 10.14309/ajg.0000000000001805. Epub 2022 May 9. PMID 35537858
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Functional Dyspepsia - Cannabidiol: Cannabidiol will be administered to participants with functional dyspepsia orally twice daily in equally divided doses starting at 2.5mg/kg per day and increasing by 2.5 to 5.0mg/kg every other day until the target dose of 20mg/kg is reached.
- Functional Dyspepsia - Placebo: Placebo will be administered to participants with functional dyspepsia orally twice daily in equally divided doses starting at 2.5mg/kg per day and increasing by 2.5 to 5.0mg/kg every other day until the target dose of 20mg/kg is reached.
- Gastroparesis - Canabidiol: Cannabidiol will be administered to participants with gastroparesis orally twice daily in equally divided doses starting at 2.5mg/kg per day and increasing by 2.5 to 5.0mg/kg every other day until the target dose of 20mg/kg is reached.
- Gastroparesis - Placebo: Placebo will be administered to participants with gastroparesis orally twice daily in equally divided doses starting at 2.5mg/kg per day and increasing by 2.5 to 5.0mg/kg every other day until the target dose of 20mg/kg is reached.
Period: Overall Study
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Started | 25 | 23 | 21 | 23
Completed | 22 | 21 | 20 | 22
Not Completed | 3 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo | Total
Number analyzed (Participants) | 25 | 23 | 21 | 23 | 92
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34.5 [22.9 to 48.1] | 35.0 [25.2 to 46.6] | 44.0 [32.0 to 56.0] | 44.0 [30.0 to 52.0] | 37.0 [24.0 to 52.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 19 | 20 | 75
  Male | 6 | 6 | 2 | 3 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 23 | 21 | 21 | 23 | 88
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 21 | 23 | 92

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying Half-time (T1/2) of Solids
Description: Subjects ingested a Technetium-99m sulfur colloid radiolabeled meal and Indium-111 absorbed on to activated charcoal particles and delivered to the colon by an oral methacrylate-coated capsule. Gastric emptying (GE t 1/2) was measured by scintigraphy and defined as the time required for 50% of the radiolabeled tracer to empty from the stomach.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Number analyzed (Participants) | 25 | 23 | 21 | 23
minutes | 128.7 [112.3 to 150.5] | 125.8 [120.2 to 142.2] | 246.4 [172.1 to 312.9] | 198.4 [148.9 to 241.3]

2. Primary Outcome: Gastric Emptying Lag Time (T-lag) of Solids
Description: Subjects ingested a Technetium-99m sulfur colloid radiolabeled meal and Indium-111 absorbed on to activated charcoal particles and delivered to the colon by an oral methacrylate-coated capsule. Gastric emptying lag time (GE t-lag) was measured by scintigraphy and defined as the amount of time the radioactive meal was in the stomach before starting to empty into the small bowel.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Number analyzed (Participants) | 25 | 23 | 21 | 23
minutes | 46.0 [34.3 to 60.0] | 52.1 [30.0 to 64.2] | 83.0 [67.5 to 128.0] | 60.8 [35.0 to 94.0]

3. Primary Outcome: Fasting Gastric Volume
Description: Gastric fasting volume was measured prior to a meal of 300 mL standardized radio-labeled Ensure drink using an intravenous injection of Technetium Tc-99m pertechnetate and noninvasive single photon emission-computed tomography (SPECT).
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Number analyzed (Participants) | 25 | 23 | 21 | 23
mL | 179.0 [161.1 to 212.0] | 214.5 [173.7 to 263.8] | 235.6 [170.8 to 319.0] | 220.3 [187.2 to 292.2]

4. Primary Outcome: Gastric Accommodation
Description: Gastric accommodation was measured 15 minutes after ingestion of 300 mL standardized radio-labeled Ensure drink using an intravenous injection of Technetium Tc-99m pertechnetate and noninvasive single photon emission-computed tomography (SPECT).
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Number analyzed (Participants) | 25 | 23 | 21 | 23
mL | 410.2 [324.9 to 451.1] | 417.5 [318.7 to 473.6] | 440.6 [392.8 to 467.8] | 415.5 [353.2 to 456.0]

5. Primary Outcome: Satiation Volume to Fullness
Description: Thirty (30) minutes after ingesting the meal of 300 mL radio-labeled Ensure drink, an additional Ensure drink was ingested at a constant rate of 30 mL/min. Participants recorded their sensations every 5 minutes using a numeric scale from 0 to 5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal, and level 5 corresponding to the MTV (maximum or unbearable fullness/satiation). Nutrient intake was stopped when subjects reach a score of 5.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Number analyzed (Participants) | 25 | 23 | 21 | 23
mL | 373.3 [373.3 to 559.9] | 622.1 [373.3 to 746.6] | 682.6 [631.2 to 826.5] | 638.2 [575.3 to 710.7]

6. Primary Outcome: Satiation Maximum Tolerated Volume (MTV)
Description: as for outcome 5
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Number analyzed (Participants) | 25 | 23 | 21 | 23
mL | 808.8 [435.8 to 995.4] | 871.0 [497.7 to 1119.8] | 1061.6 [812.7 to 1310.4] | 812.7 [688.3 to 1061.6]

7. Secondary Outcome: Weekly Global Symptom Assessment
Description: The number of functional dyspepsia participants who confirmed adequate relief of dyspepsia symptoms, based on the self-reporting question "In the past 7 days have you had adequate relief of your upper abdominal pain or discomfort?".
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo
Number analyzed (Participants) | 25 | 23
Participants | 12 | 11

8. Secondary Outcome: Mean Daily Symptom Score in Functional Dyspepsia
Description: Self-reported daily symptom diaries assessed 3 symptoms of functional dyspepsia: (1) upper abdominal pain, (2) nausea, and (3) bloating or distension. Each symptom was scored from 0-4, where 0=none, 1= very mild, 2=mild, 3=moderate, and 4=severe. The responses were averaged together to provide an overall symptom score, which ranged from 0-4, where a higher score reflects worse symptoms.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo
Number analyzed (Participants) | 25 | 23
score on a scale | 1.2 [0.9 to 2.0] | 1.1 [0.8 to 2.0]

9. Secondary Outcome: Mean Daily Epigastric Pain in Functional Dyspepsia
Description: Mean daily epigastric pain in functional dyspepsia participants as measured by the question "How much did you suffer from pain in your stomach area today?". The score is based on 5 point scale ranging from 0 (not at all) to 5 (extremely) where a higher score reflects more pain.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo
Number analyzed (Participants) | 25 | 23
score on a scale | 0.7 [0.1 to 1.3] | 0.8 [0.3 to 1.1]

10. Secondary Outcome: Quality of Life in Functional Dyspepsia
Description: The Nepean Dyspepsia Index (NDI) is used to assess functional dyspepsia quality of life. NDI scores are summarized as overall quality of life based on 5 subscales: interference, knowledge/control, eating/drinking, sleep disturbance, work/study. There are two questions per subscale for a total of 10 questions. Each question is ranked from 0-4, where 0 is 'not at all' and 4 is 'extremely'. The results from each question are added together to generate a total index score of 0 to 40. A lower score reflects no to little impact functional dyspepsia has on on quality of life while a higher score reflects significant impact functional dyspepsia has on quality of life.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo
Number analyzed (Participants) | 25 | 23
score on a scale | 4.4 [3.2 to 5.0] | 3.6 [3.0 to 4.7]

11. Secondary Outcome: Aggregate Symptom Score
Description: Postprandial symptoms of fullness, nausea, bloating, and pain were measured 30min after the satiation drink test using 100mm horizontal visual analog scales, with the words "none" and "worst ever" anchored at each end. Scores for each symptom were added to calculate the aggregate symptom score, which ranged from 0-400, where a lower score reflected mild symptoms and a higher score reflected more severe symptoms.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Number analyzed (Participants) | 25 | 23 | 21 | 23
score on a scale | 182.5 [132.5 to 253.0] | 219.0 [184.0 to 250.0] | 243.0 [234.0 to 313.0] | 264.5 [225.0 to 320.0]

12. Secondary Outcome: Overall Severity in Gastroparesis
Description: Overall severity in gastroparesis was self-measured daily by asking the question "In thinking about your gastroparesis disorder, what was the overall severity of your gastroparesis symptoms today (during the past 24 hours)"? The responses were ranked as 0 (none), 1 (mild), 2 (moderate), 3 (severe) and 4 (very severe). Scores range from 0-4, where 0 reflects little to no severity of symptoms and 4 reflects severe symptoms.
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Number analyzed (Participants) | 21 | 23
score on a scale | 1.8 [1.3 to 2.5] | 1.6 [1.2 to 3.1]

13. Secondary Outcome: Average Daily Vomiting Episodes in Gastroparesis
Description: The average daily number of vomiting episodes in gastroparesis was measured by participants self-reporting responses to the question "In the past 24 hours how many episodes of vomiting did you have?"
Time Frame: 4 weeks
Measure: Median (Inter-Quartile Range); unit: vomiting episodes/day
Arm/Group | Gastroparesis - Canabidiol | Gastroparesis - Placebo
Number analyzed (Participants) | 21 | 23
vomiting episodes/day | 0.0 [0.0 to 0.1] | 0.2 [0.0 to 0.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each subject from baseline until 30 days after the last day of study medication, for approximately two months.
Arm/Group | Functional Dyspepsia - Cannabidiol | Functional Dyspepsia - Placebo | Gastroparesis - Canabidiol | Gastroparesis - Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/23 | 0/21 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/23 | 2/21 | 0/23
Other Adverse Events (participants affected / at risk) | 11/25 | 8/23 | 19/21 | 10/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Dyspepsia - Cannabidiol (N=25) | Functional Dyspepsia - Placebo (N=23) | Gastroparesis - Canabidiol (N=21) | Gastroparesis - Placebo (N=23)
Abdominal lacerations (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendectomy (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Functional Dyspepsia - Cannabidiol (N=25) | Functional Dyspepsia - Placebo (N=23) | Gastroparesis - Canabidiol (N=21) | Gastroparesis - Placebo (N=23)
Fatigue (General disorders) | 8 (8) | 8 (8) | 4 (4) | 4 (4)
Nausea (General disorders) | 8 (8) | 8 (8) | 3 (3) | 4 (4)
Diarrhea (General disorders) | 8 (8) | 1 (1) | 12 (12) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/88/NCT03941288/Prot_SAP_001.pdf
  • Informed Consent Form (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/88/NCT03941288/ICF_000.pdf